CLINICAL TRIAL: NCT00504881
Title: An International, Randomized, Double-blind, Parallel-group, Placebo-controlled, Flexible Dose Study: Evaluation of the Safety and Efficacy of Brivaracetam in Subjects (≥ 16 to 70 Years Old) Suffering From Localization-related or Generalized Epilepsy.
Brief Title: Brivaracetam as add-on Treatment in Adolescents and Adults Suffering From Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01254; 2006-006346-34 (EudraCT Number)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo tablets administered twice a day
  Interventions: Drug: Placebo
- Brivaracetam (Experimental): A flexible dose of Brivaracetam tablets, administered twice a day, starting with a dose of 20 mg/day and could increase to 50 mg/day, 100 mg/day or 150 mg/day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Placebo — Daily oral dose of two equal intakes, morning and evening, of Placebo in a double-blinded way for the 16-week Treatment Period
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, Brivaracetam 20 mg/day or Brivaracetam 50 mg/day or Brivaracetam 100 mg/day or Brivaracetam 150 mg/day, in a double-blinded way for the 16-week Treatment Period
  Arms: Brivaracetam

SUMMARY:
This study will compare the safety and efficacy of Brivaracetam at flexible dose with Placebo in subjects suffering from Epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were aged from 16 to 70 years, inclusive. Subjects under 18 years of age were only included where legally permitted and ethically accepted
* Subjects had well-characterized localization-related Epilepsy or generalized Epilepsy according to the International League Against Epilepsy (ILAE) classification
* For subjects suffering from localization-related Epilepsy: subjects had at least 2 Partial-Onset Seizures (POSs) whether or not secondarily generalized per month during the 3 months preceding Visit 1 according to the ILAE classification
* For subjects suffering from localization-related Epilepsy: subjects had at least 4 Partial-Onset Seizures (POSs) whether or not secondarily generalized during the 4-week Baseline Period according to the ILAE classification
* For subjects suffering from generalized Epilepsy: subjects had at least 2 Type II-seizure days per month during the 3 months preceding Visit 1 according to the ILAE classification
* For subjects suffering from generalized Epilepsy: subjects had at least 4 Type II-seizure days during the 4 week Baseline Period according to the ILAE classification
* Subjects were uncontrolled while treated by 1 to 3 permitted concomitant Antiepileptic Drugs (AEDs). Vagal nerve stimulation was allowed and was not counted as a concomitant AED

Exclusion Criteria:

* For subjects who suffered from localization-related Epilepsy: history or presence of Seizures occurring only in clusters (too frequently or indistinctly separated to be reliably counted) before Visit 2 or occurring only as Type IA non-motor
* Subjects with a history or presence of Status Epilepticus during the year preceding Visit 1 or during Baseline

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (61):
- Austria (4):
  - Graz
  - Innsbrick
  - Linz
  - Vienna
- Belgium (4):
  - Bruges
  - Godinne
  - Leuven
  - Montignies-sur-Sambre
- Czechia (5):
  - Beroun
  - Brno
  - Ostrava Trebovice
  - Prague
  - Zlín
- Germany (7):
  - Berlin
  - Bernau
  - Bielefeld
  - Erlangen
  - Göttingen
  - Jena
  - München
- Hong Kong, Hong Kong
- India (6):
  - Bangalore
  - Hyderabad
  - Mumbai
  - New Delhi
  - Pune Maharashtra
  - Tirupati
- Italy (5):
  - Bari
  - Milan
  - Pavia
  - Roma
  - Siena
- Norway (5):
  - Bergen
  - Fredrikstad
  - Oslo
  - Sandvika
  - Trondheim
- Russia (5):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara
  - Yaroslavi
- Singapore, Singapore
- South Africa (4):
  - Cape Town
  - George
  - Johannesburg
  - Tygeberg
- South Korea (2):
  - Gwangju
  - Seoul
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Umeå
- Taiwan (3):
  - Taichung
  - Tainan
  - Taoyuan Hsien
- Ukraine (6):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Uzhhorod

REFERENCES:
- [Result] Kwan P, Trinka E, Van Paesschen W, Rektor I, Johnson ME, Lu S. Adjunctive brivaracetam for uncontrolled focal and generalized epilepsies: results of a phase III, double-blind, randomized, placebo-controlled, flexible-dose trial. Epilepsia. 2014 Jan;55(1):38-46. doi: 10.1111/epi.12391. Epub 2013 Oct 3. PMID 24116853
- [Result] Mukuria C, Young T, Keetharuth A, Borghs S, Brazier J. Sensitivity and responsiveness of the EQ-5D-3L in patients with uncontrolled focal seizures: an analysis of Phase III trials of adjunctive brivaracetam. Qual Life Res. 2017 Mar;26(3):749-759. doi: 10.1007/s11136-016-1483-3. Epub 2016 Dec 21. PMID 28004320
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in 15 countries. It started in October 2007 and concluded in December 2008.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS).
Period: Overall Study
Arm/Group | Placebo | Brivaracetam
Started | 121 | 359
Completed | 111 | 323
Not Completed | 10 | 36
Not completed — Lack of Efficacy | 1 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Non-Compliance | 1 | 0
Not completed — No Birth Control | 0 | 1
Not completed — Safety Visit not performed | 0 | 1
Not completed — AE, serious fatal | 0 | 1
Not completed — SAE, non-fatal | 2 | 6
Not completed — AE, non-serious non-fatal | 4 | 14
Not completed — SAE,non-fatal+AE,non-serious non-fatal | 0 | 2
Not completed — AE of unknown type | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Randomized Set (RS).
Arm/Group | Placebo | Brivaracetam | Total Title
Number analyzed (Participants) | 121 | 359 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 8
  Between 18 and 65 years | 116 | 352 | 468
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.5) | 35.6 (11.5) | 35.85 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 178 | 230
  Male | 69 | 181 | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event During the 16-week Treatment Period
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Week 2 to the end of the Treatment Period (Week 16)
Population: The Safety Population was defined as all randomized subjects who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 121 | 359
percentage of participants | 66.1 | 66.6

2. Primary Outcome: Partial Onset Seizure (Type I) Frequency Per Week Over the 16-week Treatment Period
Description: Partial (Type I) seizures can be classified into one of the following three groups:
  * Simple partial seizures
  * Complex partial seizures
  * Partial seizures evolving to generalized tonic-clonic convulsions.
  Partial Onset Seizure (POS) frequency per week over the Treatment Period (TP) was calculated as:
  (Total Type I seizures over the TP)*7/(Total number of days with no missing seizure count in the TP)
Time Frame: Baseline (Week 0) to the end of the Treatment Period (Week 16)
Population: Localization-related epilepsy Intent-To-Treat (ITT) Population (POS). The ITT Population was defined as all randomized subjects who received at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
seizures per week | 1.86 [1.00 to 3.98] | 1.74 [0.86 to 4.04]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam; ANCOVA on log-transformed partial seizure frequency per week over the treatment period, with log-transformed baseline seizure frequency per week as covariate, and including terms for treatment and stratification factors; Test type: Superiority or Other; p = 0.125, ANCOVA; Percent Reduction over Placebo = 7.3, 95% CI 2-sided [-2.2 to 15.9]

3. Secondary Outcome: Responder Rate for Partial Onset Seizures (Type I) Frequency Per Week Over the 16-week Treatment Period
Description: The responder rate was presented as the percentage of responders and non-responders. A subject is a responder, if the subject has at least 50 % reduction in Partial Onset Seizure frequency per week from Baseline to Treatment Period. Subjects with zero seizure frequency per week at Baseline were considered as non-responders.
Time Frame: Baseline (Week 0) to the end of Treatment Period (Week 16)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
percentage of participants
  Responders | 16.7 | 30.3
  Non-Responders | 83.3 | 69.7

4. Secondary Outcome: Seizure Frequency (All Seizure Types) Per Week Over the 16-week Treatment Period
Description: There are three different types of seizures:
  * Type I: Partial seizures
  * Type II: Generalized seizures
  * Type III: Unclassified epileptic seizures. All seizure frequency per week over Treatment Period (TP) was calculated as: (Total number of seizures over the TP)*7/(Total number of days with no missing seizure count in the TP)
Time Frame: Baseline (Week 0) to the end of Treatment Period (Week 16)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: number of seizures per week
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
number of seizures per week | 1.87 [1.00 to 4.59] | 1.74 [0.86 to 4.04]

5. Secondary Outcome: Percent Change From Baseline to the 16-week Treatment Period in Partial Onset Seizure (Type I) Frequency Per Week
Description: Percent change from Baseline was calculated as percent reduction by:
  (weekly seizure frequency Baseline - weekly seizure frequency Treatment)*100/(weekly seizure frequency Baseline).
  A negative value in percent Change from Baseline indicates an improvement from Baseline.
  The higher the negative values for percent change in Partial Onset Seizure (POS) frequency, the higher the improvement from Baseline.
Time Frame: Baseline (Week 0) to end of Treatment Period (Week 16)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
percent change | -18.93 [-39.05 to -7.83] | -26.92 [-55.98 to 11.44]

6. Secondary Outcome: Categorized Response From Baseline in Seizure Frequency for Partial Onset Seizure (Type I) Over the 16-week Treatment Period
Description: Subjects were classified in 1 of the following categories based on their percent reduction from Baseline to Treatment Period in Partial Onset Seizure (POS) frequency per week: <-25 %, -25 % to <25 %, 25 % to <50 %, 50 % to <75 %, 75 % to <100 %, and 100 %.
  Subjects having zero for Baseline seizure frequency per week were classified in the <-25 % category.
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
percentage of participants
  <- 25 % | 14.8 | 18.3
  -25 % to < 25 % | 44.4 | 29.1
  25 % to < 50 % | 24.1 | 22.3
  50 % to < 75 % | 13.9 | 17.0
  75 % to < 100 % | 2.8 | 11.8
  100 % | 0 | 1.5

7. Secondary Outcome: Seizure Freedom Rate (All Seizure Types) Over the 16-week Treatment Period
Description: Subjects were considered seizure free if their seizure counts for every day over the Treatment Period (TP) was zero and if they did not discontinue before the end of the TP. Seizure freedom rate was calculated as:
  (total number of seizure - free subjects in treatment group during TP)/(total number of evaluable Intent-To-Treat (ITT) subjects in treatment group)
Time Frame: Baseline (Week 0) to the end of Treatment Period (Week 16)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
percentage of participants
  Seizure-free | 0 | 1.5
  No Seizure but non-completer | 0 | 0
  Not Seizure free | 100.0 | 98.5

8. Secondary Outcome: Reduction of Type IC/Type I Seizure Frequency Ratio From Baseline to the 16-week Treatment Period
Description: The type IC/Type I seizure frequency ratio is represented by the percentage of subjects having a reduction in the ratio of Type IC seizure frequency over Type IA, IB, and IC seizure frequency from Baseline to Treatment Period.
Time Frame: Baseline to 16-week Treatment Period
Population: The Intention-to-treat (ITT) population was defined as all randomized subjects who received at least 1 dose of study medication.
  Type IC Population consists of those subjects with at least one Type IC seizure during the Baseline period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 35 | 94
percentage of participants | 54.3 | 47.9

9. Secondary Outcome: Time to First Type I Seizure During the 16-week Treatment Period
Description: Time to first Type I seizure during the 16-week Treatment Period was measured in days.
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
days | 3 [2 to 4] | 4 [4 to 5]

10. Secondary Outcome: Time to Fifth Type I Seizure During the 16-week Treatment Period
Description: Time to fifth Type I seizure during the 16-week Treatment Period was measured in days.
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
days | 14 [11 to 19] | 18 [16 to 21]

11. Secondary Outcome: Time to Tenth Type I Seizure During Treatment Period
Description: Time to tenth Type I seizure during the 16-week Treatment Period was measured in days.
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 323
days | 36 [23 to 44] | 38 [31 to 43]

12. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Total Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: The Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) is an adaptation of the original QOLIE-31 instrument that includes 30 items grouped into 7 multi-item subscales: Seizure Worry (5 items), Overall Quality of Life (2 items), Emotional Well-being (5 items), Energy/Fatigue (4 items), Cognitive Functioning (6 items), Medication Effects (3 items) and Daily Activities/Social Functioning (5 items), and a Health Status item. In addition to the 31 items of the QOLIE-31, the QOLIE-31-P contains 7 items asking the subjects to rate the degree of 'distress' related to the topic of each subscale (ie, distress items). The QOLIE-31-P also contains an item asking about the relative importance of each subscale topic (ie, prioritization item). The subscale scores, the total score and the Health Status item score were calculated according to the scoring algorithm defined by the author with scores ranging from 0 to 100 and higher scores indicating better function.
Time Frame: Baseline to 16-week Treatment Period
Population: Localization-related epilepsy Intent-To-Treat (ITT) Population (POS). The ITT Population was defined as all randomized subjects who received at least 1 dose of study medication.
  Only subjects who are not mentally impaired were to complete the QOLIE-31-P. Only subjects having values at baseline and at the considered visit are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 98 | 284
units on a scale | 3.04 (12.58) | 4.22 (13.73)

13. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Seizure Worry Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 291
units on a scale | 4.66 (23.23) | 10.29 (21.99)

14. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Daily Activities / Social Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 290
units on a scale | 5.61 (21.87) | 2.66 (23.48)

15. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Hospital Anxiety Score
Description: The Hospital Anxiety and Depression Scale (HADS) was used to evaluate Anxiety and Depression. The HADS was developed as a self-administered scale to assess the presence and severity of Anxiety and Depression. It consists of 14 items that are scored on a 4-point severity scale ranging from 0 to 3. A score per dimension was calculated with each score ranging from 0 to 21 (higher scores indicating greater problems). A negative value in change from Baseline indicates an improvement from Baseline.
Time Frame: Baseline to 16-week Treatment Period
Population: Localization-related epilepsy Intent-To-Treat (ITT) Population (POS). The ITT Population was defined as all randomized subjects who received at least 1 dose of study medication.
  Only subjects who are not mentally impaired were to complete the HADS. Only subjects having values at baseline ans at the considered visit are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 97 | 286
units on a scale | -0.57 (3.35) | -0.85 (3.62)

16. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Hospital Depression Score
Description: The Hospital Anxiety and Depression Scale (HADS) was used to evaluate Anxiety and Depression.The HADS was developed as a self-administered scale to assess the presence and severity of Anxiety and Depression. It consists of 14 items that are scored on a 4-point severity scale ranging from 0 to 3. A score per dimension was calculated with each score ranging from 0 to 21 (higher scores indicating greater problems). A negative value in change from Baseline indicates an improvement from Baseline.
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 97 | 285
units on a scale | 0.30 (3.08) | -0.41 (3.54)

17. Secondary Outcome: Patient's Global Evaluation Scale (P-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: The Patient's Global Evaluation Scale (P-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1= Marked worsening to 7= Marked improvement) with the start of the study medication as the reference time point. The subject completed it by answering to the following: 'Overall, has there been a change in your seizures since the start of the study medication?'
Time Frame: Baseline to last visit or early discontinuation visit in the 16-week Treatment Period
Population: Localization-related epilepsy Intent-To-Treat (ITT) Population (POS). The ITT Population was defined as all randomized subjects who received at least 1 dose of study medication.
  Evaluable subjects are subjects who completed the GES at last treatment period visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 282
units on a scale | 4.73 (1.37) | 5.07 (1.36)

18. Secondary Outcome: Investigator's Global Evaluation Scale (I-GES) Evaluated at Last Visit or Early Discontinuation Visit
Description: The Investigator's Global Evaluation Scale (I-GES) is a global assessment of the disease evolution which was performed using a seven-point scale (1= Marked worsening to 7= Marked improvement) with the start of the study medication as the reference time point. The Investigator completed it by answering to the following: 'Assess the overall change in the severity of patient's illness, compared to start of study medication.'
Time Frame: Baseline to Last Visit or Early Discontinuation Visit in the 16-week Treatment Period
Population: Localization-related epilepsy Intent-To-Treat (ITT) Population (POS). The ITT Population was defined as all randomized subjects who received at least 1 dose of study medication.
  Evaluable subjects are subjects for whom the GES was completed by the investigator at last treatment period visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 108 | 319
units on a scale | 4.79 (1.14) | 5.00 (1.22)

19. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Energy/Fatigue Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 286
units on a scale | 2.98 (18.00) | 3.34 (19.06)

20. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Emotional Well-being Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 287
units on a scale | 1.97 (19.29) | 2.84 (18.07)

21. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Cognitive Functioning Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 290
units on a scale | 2.28 (19.88) | 5.51 (18.55)

22. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Overall Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 98 | 291
units on a scale | -0.48 (17.40) | 4.08 (19.23)

23. Secondary Outcome: Change From Baseline to the 16-week Treatment Period in Medication Effects Patient Weighted Quality of Life in Epilepsy Inventory-Form 31 (QOLIE-31-P) Score
Description: as for outcome 12
Time Frame: Baseline to 16-week Treatment Period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Brivaracetam
Number analyzed (Participants) | 99 | 290
units on a scale | 2.83 (27.21) | -0.24 (25.84)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 24 weeks from Visit 1 (Week -4) to the Safety Visit (Week 20).
Description: Adverse Events (AEs) refer to the Safety Population, including all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Placebo | Brivaracetam
Serious Adverse Events (participants affected / at risk) | 9/121 | 20/359
Other Adverse Events (participants affected / at risk) | 40/121 | 139/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=121) | Brivaracetam (N=359)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diabetis mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Postictal state (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 7 (9)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Drug toxity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=121) | Brivaracetam (N=359)
Nasopharyngitis (Infections and infestations) | 8 (10) | 14 (16)
Nausea (Gastrointestinal disorders) | 11 (14) | 20 (26)
Fatigue (General disorders) | 5 (5) | 27 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 11 (11)
Dizziness (Nervous system disorders) | 7 (9) | 31 (36)
Headache (Nervous system disorders) | 24 (45) | 52 (79)
Somnolence (Nervous system disorders) | 5 (7) | 40 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days